CLINICAL TRIAL: NCT06235125
Title: A Pilot Study of Near-Infrared Imaging Using the Novel Imaging Agent Cytalux for Adolescent Patients With Metastatic Osteosarcoma Undergoing Pulmonary Metastasectomy
Brief Title: Safety and Feasibility of Intraoperative Visualization With Cytalux in Children
Acronym: Cytalux
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: On Target Laboratories, LLC (Industry)
Responsible Party: Principal Investigator, Timothy Lautz, Director of Pediatric Surgical Oncology, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023-6263
Record Dates: First submitted 2024-01-06; First posted 2024-01-31 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Osteosarcoma; Pulmonary Metastasis; Fluorescence; Metastatic Sarcoma; Pediatrics
MeSH Terms: conditions — Osteosarcoma; Sarcoma | interventions — Pafolacianine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cytalux with Near Infrared Imaging (Experimental): All participants will receive Cytalux and undergo near infrared imaging.
  Interventions: Drug: Cytalux

INTERVENTIONS:
Drug: Cytalux — Folate analog ligand conjugated with an indole cyanine-like green dye as a solution in vials containing 3 mL at 2 mg/mL
  Other Names: Pafolacianine injection; OTL38 injection

SUMMARY:
Pediatric subjects aged 6-17 with biopsy confirmed cancer and imaging findings suspicious for pulmonary metastatic disease scheduled to undergo pulmonary metastasectomy via and open or minimally invasive approach.

DETAILED DESCRIPTION:
Pulmonary metastasectomy, or surgery to remove cancer which has spread to the lungs, plays a key role in the treatment of children with metastatic solid tumors. Fluorescence-guided surgery (FGS) has been shown to be a promising technique to highlight cancer cells and enable real-time surgical guidance (Stummer 2006, Hernot 2019, Goldstein 2021). Current techniques for fluorescence-guided surgery rely on indocyanine green (ICG), a non-specific fluorescent molecular agent which tends to accumulate in cancer cells because of increased angiogenesis and decreased lymphatic clearance. Molecular agents targeted to tumor-specific receptors offer the hope of increased sensitivity and specificity for detecting even very small metastatic nodules, and thus enhancing surgical clearance of disease.

Many of the tumors which metastasize to the lung are known to express the folate receptor and may therefore benefit from utilizing the tumor imaging agent CYTALUX (pafolacianine). CYTALUX (Pafolacianine) as a diagnostic tool during cancer resection has already been investigated in adults (approved NDA 214907), and no age-specific differences are expected in the pediatric population. Findings from the ELUCIDATE trial in adults demonstrated that intraoperative molecular imaging with CYTALUX (pafolacianine) improves surgical outcomes by identifying occult tumors and close surgical margins and it therefore gained FDA approval for adults with cancer in the lung (both primary and metastatic) as an adjunct with near infrared (NIR) imaging for detection of disease during surgery. We anticipate that this agent will have similar safety and efficacy in children and to similarly demonstrate applicable for all types of metastatic tumors.

This is a pilot study in pediatric subjects aged 6-17 with biopsy confirmed cancer and imaging findings suspicious for pulmonary metastatic disease scheduled to undergo pulmonary metastasectomy via an open or minimally invasive approach.

In the proposed study, subjects and their parents or guardians will give informed consent prior to commencement of any study procedures. Subjects will be dosed with 0.025 mg/kg CYTALUX (pafolacianine) injection intravenously from 4 hours to up to 24 hours prior to surgery. Subjects will be considered evaluable if they are exposed to study drug and/or NIR fluorescent light imaging. During surgery, all subjects will first undergo evaluation by normal surgical techniques (white light, palpation, and/or other localization techniques) and all suspicious nodules and lesions identified under standard surgical approach will be recorded as such. Following standard surgical assessment, subjects will undergo assessment with NIR fluorescent light imaging prior to and after resection.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 6-17 years of age at the time of study enrollment
2. Willingness of research participant or legal guardian/representative to give written informed consent
3. Willingness of patients (subjects) age 12-17 to provide written adolescent assent
4. Patient weight greater than or equal to 20 kg
5. Histologically confirmed diagnosis of osteosarcoma, synovial sarcoma, hepatoblastoma, rhabdomyosarcoma, Ewing sarcoma, Wilms tumor or other non-rhabdomyosarcoma soft tissue sarcoma
6. Imaging findings highly suspicious for pulmonary metastatic disease based on CT, PET-CT or other imaging and warranting pulmonary surgery based on the judgment of the treating team. At least one nodule ≥4mm measured by preoperative imaging.
7. Female (assigned female at birth) participant is not pregnant and agrees to an acceptable form of contraception from the time of consent through 30 days after study intervention. Confirmed abstinence is an acceptable form of contraception.
8. Female (assigned female at birth) participant must agree to not donate ova from time of consent until 30 days after study intervention
9. Male (assigned male at birth) participant must agree to not donate sperm from time of consent until 30 days after study intervention.

Exclusion Criteria:

1. Any medical condition that in the opinion of the investigators could potentially jeopardize the safety of the subject
2. History of anaphylactic reactions to products containing indocyanine green for near infrared imaging. Subjects with a medical history of 'idiopathic anaphylaxis' will also be excluded.
3. History of allergy to any of the components of CYTALUX™ (PAFOLACIANINE) INJECTION
4. Presence of any psychological, familial, sociological condition or geographical challenges potentially hampering compliance with the study protocol or follow-up schedule
5. Impaired renal function defined as eGFR< 50 mL/min/1.73m2
6. Impaired liver function defined as values > 3x the upper limit of normal (ULN) for alanine aminotransferase (ALT) or aspartate aminotransferase (AST), alkaline phosphatase (ALP), or >2x ULN for total bilirubin except in subjects with Gilbert's syndrome.
7. Patient unable or unwilling to discontinue folate, folic acid, or folate-containing supplements 48 hours before study drug administration
8. History of drug-related serious adverse event with prior Cytalux administration will be an exclusion for re-enrollment for contralateral surgery (see section 5.7).
9. Participants will be excluded if their 12th or 18th birthday would occur during study participation
10. Male sex at birth and commitment to acceptable form of contraception from time of consent through 30 days after study intervention with confirmed abstinence as an acceptable form of contraception as an inclusion criterion.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2024-04-08 (Actual); Primary Completion 2026-01-20 (Estimated); Study Completion 2026-01-20 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of Near-infrared (NIR) imaging after pafolacianine injection for metastatic nodule identification | 1 day
  In children and adolescents with histologically-confirmed cancer undergoing pulmonary surgery for suspected metastases, each excised pulmonary lesion will be classified by the surgeon as positive or negative on NIR imaging after administration CYTALUX™ (PAFOLACIANINE) and then subjected to routine histologic examination. Sensitivity will be assessed as the fraction of histologically-confirmed metastatic nodules which demonstrated positive NIR fluorescence.
False-Positive Rate of Near-infrared (NIR) imaging after pafolacianine injection for metastatic nodule identification | 1 day
  In children and adolescents with histologically-confirmed cancer undergoing pulmonary surgery for suspected metastases, each excised pulmonary lesion will be classified by the surgeon as positive or negative on NIR imaging after administration CYTALUX™ (PAFOLACIANINE) and then subjected to routine histologic examination. The false positive rate will be assessed as the fraction of NIR-positive nodules that have no viable malignancy on histologic examination.

SECONDARY OUTCOMES:
Detection of occult metastatic lesion(s) with Near-infrared (NIR) imaging after pafolacianine injection | 1 day
  The proportion of subjects with one or more NIR-positive lesion(s), not detected under normal light and/or palpation, and subsequently determined on histologic evaluation to contain viable metastatic tumor
Number of patients with treatment-emergent adverse events (TEAEs) | 30 days
  Adverse events (AEs) will be coded using MedDRA. An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. A TEAE is defined as an AE observed after administration of the study intervention and up to the follow-up period. The number of TEAEs will be collected to asses the safety and tolerability of single intravenous infusions/injection of CYTALUX™ (PAFOLACIANINE) INJECTION in children and adolescents

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Lautz, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H. Lurie Children's Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sarkaria IS, Martin LW, Rice DC, Blackmon SH, Slade HB, Singhal S; ELUCIDATE Study Group. Pafolacianine for intraoperative molecular imaging of cancer in the lung: The ELUCIDATE trial. J Thorac Cardiovasc Surg. 2023 Dec;166(6):e468-e478. doi: 10.1016/j.jtcvs.2023.02.025. Epub 2023 Mar 3. PMID 37019717